CLINICAL TRIAL: NCT00062400
Title: A Survey of the Breast International Group (B.I.G.) to Assess the Attitude of Patients Aged Less Than 35 Years, With Early Breast Cancer, Toward the Risk of Loss of Fertility Related to Adjuvant Therapies
Brief Title: Assessing Women's Attitudes About the Risk of Infertility Related to Adjuvant Therapy for Early Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: German Adjuvant Breast Cancer Group (Other); ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-10002; EORTC-10002; BIG-3-98; IBCSG-29-03
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer; Psychosocial Effects of Cancer and Its Treatment; Sexual Dysfunction and Infertility; Sexuality and Reproductive Issues
Keywords: sexual dysfunction and infertility; sexuality and reproductive issues; psychosocial effects of cancer and its treatment; stage II breast cancer; stage IA breast cancer; stage IB breast cancer
MeSH Terms: conditions — Breast Neoplasms; Sexual Dysfunction, Physiological; Infertility; Sexuality | interventions — Psychiatric Rehabilitation

INTERVENTIONS:
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Adjuvant therapy given after surgery for early breast cancer may cause infertility. Assessing young women's attitudes and feelings about the risk of infertility may help improve the ability to plan effective treatment.

PURPOSE: This clinical trial is studying young women's attitudes and feelings about the risk of infertility related to adjuvant therapy for stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the attitude toward the risk of infertility related to adjuvant therapy in women with early breast cancer.
* Correlate, if possible, the patient's attitude with the fact that the patient already has children or the time interval between the date of breast cancer diagnosis and the date of study participation.

OUTLINE: This is a multicenter study.

Patients complete a questionnaire administered by a nontreating physician.

PROJECTED ACCRUAL: A total of 385 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed prior or current diagnosis of breast cancer

  * Stage I or II
  * No relapsed disease
* No evidence of infertility

  * Regular menses or regular hormonal contraception use for the past 3 months
* Hormonal status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 35 and under at diagnosis

Sex

* Female

Menopausal status

* Premenopausal

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No psychological, familial, sociological, or geographical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* Not specified

Surgery

* Not specified

Max Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 385 (Estimated)
Dates: Start 2003-05; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Patients who would agree to have chemotherapy if it reduces their chances of having children as assessed by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Zora Neskovic-Konstantinovic, Study Chair — Institute Of Oncology & Radiology, Belgrade, Serbia
Locations (27):
- Belgium (4):
  - Institut Jules Bordet, Brussels
  - Centre Hospitalier Etterbeek Ixelles, Brussels
  - CHU Liege - Domaine Universitaire du Sart Tilman, Liège
  - Algemeen Ziekenhuis Sint-Augustinus, Wilrijk
- Chile (3):
  - Instituto de Radiomedicina, Santiago
  - Clinica Alemana, Santiago
  - Hospital Militar, Santiago
- University Hospital Rebro, Zagreb, Croatia
- Germany (2):
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Universitatsklinikum Heidelberg, Heidelberg
- Italy (4):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Azienda Istituti Ospitalieri, Cremona
  - Ospedale Alessandro Manzoni, Lecco
  - European Institute of Oncology, Milan
- American University of Beirut Medical Center, Beirut, Lebanon
- Netherlands (2):
  - Academisch Medisch Centrum at University of Amsterdam, Amsterdam
  - Arnhems Radiotherapeutisch Instituut, Arnhem
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru
- Medical University of Gdansk, Gdansk, Poland
- Instituto Portugues de Oncologia de Francisco Gentil - Centro Regional de Oncologia de Lisboa, SA, Lisbon, Portugal
- Institute of Oncology and Radiology of Serbia, Belgrade, Serbia
- Groote Schuur Hospital, Cape Town, South Africa
- Switzerland (3):
  - Inselspital Bern, Bern
  - Ospedale Beata Vergine, Mendrisio
  - Kantonsspital - St. Gallen, Sankt Gallen
- Marmara University Hospital, Istanbul, Turkey (Türkiye)
- Western Infirmary, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Result] Neskovic-Konstantinovic Z, Gomez H, Senkus-Konefka E, et al.: A Breast International Group survey of young breast cancer patients attitudes towards the risk of loss of fertility related to adjuvant therapies: EORTC protocol 10002 - BIG 3-98. [Abstract] 31st Annual San Antonio Breast Cancer Symposium, December 10-14, 2008, San Antonio, Texas. A-3106, 2008.